CLINICAL TRIAL: NCT06613776
Title: Evaluation of the Effect of Antibiotic Prophylaxis on Inflammatory Factor in Salivary Samples After Third Molars Surgery
Brief Title: Evaluation of the Effect of Antibiotic Prophylaxis (2g Amoxicillin One Hour Before Surgery) on an Inflammatory Factor (PGE2) in Salivary Samples After Third Molars Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Carlos Pérez-Albacete Martínez, Prof. Dr., Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CE032315
Record Dates: First submitted 2024-09-20; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Third Molar Extraction Surgery; Antibiotic Prophylaxis; Amoxicillin
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Antibiotic) (Experimental): 4 amoxicillin 500 mg capsules (2 grams)
  Interventions: Drug: Amoxicillin
- Control group (Placebo) (Placebo Comparator): 4 empty amoxicillin 500mg capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin — 4 capsules of amoxicillin 500mg, 2 grams in total, one hour before surgery
  Arms: intervention group (Antibiotic)
Drug: Placebo — 4 empty capsules of amoxicillin 500mg (placebo), one hour before surgery
  Arms: Control group (Placebo)

SUMMARY:
This clinical trial aims to evaluate the impact of antibiotics on inflammation and pain in patients who have undergone mandibular third molar surgery. The primary research questions are:

1. Do antibiotics reduce pain following third molar surgery?
2. Do antibiotics influence facial swelling and the patient's ability to open their mouth?
3. Do antibiotics affect the levels of a specific inflammatory marker in saliva post-surgery?

Participants will be randomly assigned to receive either antibiotic capsules or placebo capsules. The study will include the following procedures:

Medication: Participants will take four capsules (either antibiotics or placebo) as part of their standard surgical care.

Saliva Samples: Saliva samples will be collected at three time points: before surgery, 24 hours after surgery, and 7 days post-surgery.

Measurements: Facial swelling and mouth opening will be assessed by the investigator at each time point.

By comparing the outcomes between the antibiotic and placebo groups, researchers aim to determine the effectiveness of antibiotics in managing post-surgical inflammation and pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people (ASA I & II)
* Older than 18 years
* No history of viral or microbial diseases during the last four months
* No history of allergic reaction to penicillin-class antibiotics or other drugs that will be used during the research
* No history of anti-inflammatory or contraceptive drugs use during the last month
* Not being in pregnancy or nursing period for women
* Having at least one unerupted mandibular wisdom tooth needs surgical intervention

Exclusion Criteria:

* History of dental pain, inflammation, or abscess during the last month
* thyroid hormone therapy
* unwillingness to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Pain reported by patients | From the first visit immediately after surgery to the last visit, 6 days.
  Pain levels are assessed using a Visual Analog Scale (VAS) and a 10-point scale at several intervals: immediately after surgery, at 6 hours, 12 hours, and 24 hours post-surgery, and daily at 17:00 until the 6th day post-surgery. On this scale, 0 indicates no pain, while 10 represents the worst pain the patient has ever experienced.

SECONDARY OUTCOMES:
Maximum mouth opening change | From the initial visit before surgery to the final visit 7 days post-surgery, at 7 days
  Using a metal ruler, measure the maximum distance (in millimeters) between the incisal edge of the maxillary incisor and the lower incisor. The researcher will evaluate the maximum mouth opening at four time points: before surgery, immediately after surgery, 24 hours post-surgery, and 7 days post-surgery. The change in maximum mouth opening will be calculated by comparing the pre-surgery measurement with each subsequent measurement. Fewer changes are favorable.
Facial swelling | From the day of surgery to the last visit, at 7 days
  Facial swelling is assessed using a tape-measuring method. The patient sits upright at a 90˚ angle with their mandible at rest. Three facial measurements are taken:
  Line A: Distance from the tragus to the corner of the mouth Line B: Distance from the tragus to the soft tissue pogonion Line C: Distance from the outer corner of the eye to the angle of the mandible The facial measurement formula is ((A + B + C) / 3). Facial swelling (%) is calculated as ([postoperative measurement on T2 - preoperative measurement]/preoperative measurement) *100 Less facial swelling is favorable.

CONTACTS AND LOCATIONS:
Locations (1):
- UCAM dental, Clinica odontologica universitaria, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) underlying the results in a publication will be shared, ensuring the protection of patients' personal information.
Supporting Information: Study Protocol, ICF
Time Frame: Data sharing will begin with the publication of results and will have no end date.

REFERENCES:
- [Background] Torof E, Morrissey H, Ball PA. The Role of Antibiotic Use in Third Molar Tooth Extractions: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2023 Feb 21;59(3):422. doi: 10.3390/medicina59030422. PMID 36984426
- [Background] Mehra P, Reebye U, Nadershah M, Cottrell D. Efficacy of anti-inflammatory drugs in third molar surgery: a randomized clinical trial. Int J Oral Maxillofac Surg. 2013 Jul;42(7):835-42. doi: 10.1016/j.ijom.2013.02.017. Epub 2013 Mar 25. PMID 23535007